CLINICAL TRIAL: NCT03738969
Title: Longitudinal Study of Different Surgical Approaches in Chinese Patients of Cervical Cancer
Brief Title: Longitudinal Study of Different Surgical Approaches in Chinese Patients of Uterine Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: SACCC
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Uterine Cervical Neoplasms; Laparotomy; Laparoscopy; Survival; Mortality; Recurrence
MeSH Terms: conditions — Uterine Cervical Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Laparotomy group: Patients in this group accepted laparotomic radical hysterectomy for cervical cancer.
  Interventions: Procedure: Laparotomic radical hysterectomy
- Laparoscopy group: Patients in this group accepted laparoscopic or robotic radical hysterectomy for cervical cancer.
  Interventions: Procedure: Laparoscopic radical hysterectomy

INTERVENTIONS:
Procedure: Laparotomic radical hysterectomy — Radical hysterectomy applied by laparotomy
  Groups: Laparotomy group
Procedure: Laparoscopic radical hysterectomy — Radical hysterectomy applied by laparoscopic
  Groups: Laparoscopy group

SUMMARY:
This multi-center longitudinal study aims to compare the survival outcomes (including overall survival, progression-free survival and disease-free survival between uterine cervical patients receiving different surgical routes (vaginal, laparotomy and laparoscopy), which is the primary study objective. All clinical and pathological data would be retracted from case reviews, and all survival data would be reached by clinic, telephone and mail follow-up. This study also would analyze the impact on survival outcomes of other factors, including nerve-sparing techniques, neoadjuvant chemotherapy, neoadjuvant radiotherapy and infection of human papillomavirus. The predictive effects of different following protocol and imaging plans will be also compared. Last, the influences of surgical routes on the fertility outcomes (pregnancy and its complications) and the ovarian reserve are important secondary study objectives.

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmed as uterine cervical cancer
* Having definite clinical information
* Having received radical hysterectomy or trachelectomy

Exclusion Criteria:

* Not satisfying any of the inclusion criteria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients pathological confirmed as uterine cervival cancer and receiving radical hysterectomy or trachelectomy would been included.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2018-11-10 (Actual); Primary Completion 2022-12-23 (Estimated); Study Completion 2023-12-23 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Five years
  Length of time during and after the treatment of cervical cancer, that a patient lives with the disease but it does not get worse

SECONDARY OUTCOMES:
Overall survival | Five years
  The length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive. In a clinical trial, measuring the overall survival is one way to see how well a new treatment works.
Disease-free survival | Five years
  In cancer, the length of time after primary treatment for a cancer ends that the patient survives without any signs or symptoms of that cancer. In a clinical trial, measuring the disease-free survival is one way to see how well a new treatment works.

OTHER OUTCOMES:
Pregnancy rate | Five years
  Proportion of patients who have been pregnant after the fertility-preserving radical trachelectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All the data will be available to all researchers on the public websites
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Derived] Chao X, Wu M, Ma S, Tan X, Zhong S, Song X, Li L. Efficacy of different surgical approaches on survival outcomes in patients with early-stage cervical cancer: protocol for a multicentre longitudinal study in China. BMJ Open. 2020 Aug 20;10(8):e038020. doi: 10.1136/bmjopen-2020-038020. PMID 32819996